CLINICAL TRIAL: NCT06877351
Title: Oral Amoxicillin Compared to Penicillin G Benzathine for the Treatment of Acquired Syphilis in Pediatric Population: Prospective, Open-label, Non-inferiority, Multicenter Trial
Brief Title: Oral Amoxicillin Compared to Penicillin G Benzathine for the Treatment of Acquired Syphilis.
Acronym: AMOXSYP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Responsible Party: Principal Investigator, GUILLERMO FERNANDO MOSCATELLI, Prof Dr Guillermo F Moscatelli, Hospital de Niños R. Gutierrez de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13246
Record Dates: First submitted 2025-03-05; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-12

CONDITIONS: Syphilis Acquired
Keywords: penicillin alternatives; non-inferiority study; treponema pallidum; children; adolescents; oral amoxicillin
MeSH Terms: conditions — Treponemal Infections | interventions — Amoxicillin; Penicillin G

STUDY DESIGN:
Intervention Model Description: Randomized, phase III, multicenter, prospective, open-label, non-inferiority clinical trial.
Masking Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amoxicillin (Experimental): Amoxicillin: Administered orally at a dosage of 40-50 mg/kg/day, divided into three doses. The treatment duration is 14 days for early syphilis and 21 days for late syphilis or syphilis of unknown duration. The maximum dose is 500 mg every 8 hours.
  Interventions: Drug: Amoxicillin
- Intramuscular Penicillin G Benzathine: (Active Comparator): Intramuscular Penicillin G Benzathine: Administered as a single dose of 50,000 IU/kg for early syphilis, and as three consecutive weekly doses for late syphilis or syphilis of unknown duration. The maximum dose is 2,400,000 IU per dose.
  Interventions: Drug: Penicillin G, Benzathine

INTERVENTIONS:
Drug: Amoxicillin — Participants randomized to the intervention group will receive oral amoxicillin at a dose of 40-50 mg/kg/day (maximum 1500 mg/day), administered in three doses daily for 14 days for early syphilis and 21 days for late syphilis or syphilis of unknown duration.
  Arms: Amoxicillin
Drug: Penicillin G, Benzathine — Participants randomized to the control group will receive intramuscular procaine benzathine penicillin (PGB) at a dose of 50,000 IU/kg (maximum 2,400,000 IU/day), administered as a single dose for early syphilis and as three consecutive weekly doses for late syphilis or syphilis of unknown duration.
  Arms: Intramuscular Penicillin G Benzathine:

SUMMARY:
The goal of this clinical trial is to learn if oral amoxicillin has comparable therapeutic response than penicillin G benzathine for the treatment of acquired pediatric syphilis. It will also learn about the adverse events and biomarkers of therapeutic response associated with oral amoxicillin. The main questions it aims to answer are:

* Does comparable therapeutic response oral amoxicillin to penicillin G benzathine in the treatment of acquired pediatric syphilis?
* Does adequate serologic response to treatment participants with syphilis when taking oral amoxicillin? Researchers will compare oral amoxicillin to intramuscular procaine benzathine penicillin to see if oral amoxicillin works similar to treat acquired pediatric syphilis.

Participants will:

* Take 40-50mg/kg oral amoxicillin every day for 14 to 21 days or an intramuscular procaine benzathine penicillin injection at a dose of 50,000 IU/kg per week for one to three weeks.
* Follow-up visits every two months after treatment until a one-year follow-up is completed.
* Keep a diary of their symptoms and the number of times they take the medications

DETAILED DESCRIPTION:
A randomized, phase III, multicenter, prospective, open-label, non-inferiority clinical trial in pediatric outpatients with a diagnosis of acquired syphilis has been designed in order to compare oral amoxicillin against penicillin G benzathine for the treatment of pediatric syphilis. The primary hypothesis of this study is that oral amoxicillin is non-inferior to the standard treatment of intramuscular procaine benzathine penicillin (PGB) for the treatment of syphilis.

The primary objective of this study is to evaluate the noninferiority of oral amoxicillin compared to intramuscular PGB in treating primary, secondary, or early latent acquired syphilis in a pediatric population. The secondary outcome is to study adverse events and molecular biomarkers of therapeutic response by real-time PCR (qPCR) in both treatment arms.

Diagnostic Criteria:

Diagnosis is based on the presence of lesions compatible with syphilis, accompanied by positive results on both non-treponemal tests (VDRL/RPR) and treponemal tests (rapid strip, ELISA, or chemiluminescence).

* Primary Syphilis: Characterized by an erosion or ulceration at the site of inoculation (e.g., penis, vulva, vagina, cervix, anus, mouth). This is referred to as a "hard chancre," typically single, painless, with a hardened base and a clean ulcerated bottom.
* Secondary Syphilis: Manifested by cutaneous or mucosal lesions, which may include:

  * Erythematous Lesions: Syphilitic roseola.
  * Papular Lesions: Papular syphilids.
  * Pigmented Lesions: Nigricans and leuko-pigmented syphilids.
  * Mucosal Syphilids: Located in the mouth, larynx, pharynx, and anogenital mucosa, including erythematous, opaline, and "mown meadow" syphilids.
  * Condylomata Planaris: Papulohypertrophic, papulovegetating, or erosive papules.
  * Additional Symptoms: Alopecia, onychosis, and syphilitic paronychia.

Demographic, epidemiological, and clinical data, including information on concomitant medications, will be collected at baseline. A physical examination and comprehensive clinical evaluation will be conducted for all subjects following standard clinical practices.

Diagnostic studies will be performed in accordance with national and international standards for the diagnosis of primary and secondary syphilis. These include:

* Non-treponemal Serological Tests: For initial screening of syphilis.
* Treponemal Serological Tests: For confirmation of syphilis.
* Quantitative PCR (qPCR) Assays: To analyze whole blood samples and swabs from skin lesions, mucous membranes, and secretions.

A venous blood sample of 2 ml will be collected at diagnosis and subsequently at 2, 4, 6, 12 (endpoint), and 24 months post-treatment to evaluate the serological curve and perform molecular biology analyses

Control laboratory tests will be conducted prior to treatment and at the end of treatment (14 days post-initiation) and will include:

* Blood Count
* Hepatogram: Includes GOT, GPT, total and direct bilirubin
* Renal Function Tests: Includes urea and plasma creatinine
* Urinalysis: Single sample

Given the well-documented safety profiles of both amoxicillin and procaine benzathine penicillin (PGB), it is anticipated that no significant adverse events will occur in the treated population. Nonetheless, all participants will undergo a clinical evaluation one week after the initiation of treatment to assess any medication-related adverse events and to ensure treatment compliance.

Following this initial evaluation, participants will be contacted via telephone every two weeks until week 8 to monitor additional safety outcomes, clinical responses, and the use of concomitant medications.

Additional visits will be scheduled as needed during follow-up for patients who exhibit clinical nonresponse (persistence or worsening of lesions) within 8 weeks after the initiation of treatment, or for those who experience clinical recurrence at any point during follow-up. During these visits, epidemiological and clinical information will be gathered, and a comprehensive physical examination will be conducted. Blood samples will be collected for serological testing, and swabs will be taken from any existing lesions for further analysis.

qPCR Assays: DNA extraction will be performed using commercial columns (Qiagen, USA). Detection of Treponema pallidum pallidum (TPA) DNA will be accomplished with primers that amplify sequences from the target genes tpp47 and polA. The detection will use TaqMan probes labeled with the FAM fluorophore (Invitrogen, USA) on the CFX96 system (Bio-Rad). The human RNase P gene will serve as an internal control for the assay, while heat-killed TPA samples provided by the Centers for Disease Control and Prevention (CDC, USA) will be used as standards.

Treatment:

* Amoxicillin: Administered orally at a dosage of 40-50 mg/kg/day, divided into three doses. The treatment duration is 14 days for early syphilis and 21 days for late syphilis or syphilis of unknown duration. The maximum dose is 500 mg every 8 hours.
* Intramuscular Penicillin G Benzathine: Administered as a single dose of 50,000 IU/kg for early syphilis, and as three consecutive weekly doses for late syphilis or syphilis of unknown duration. The maximum dose is 2,400,000 IU per dose.

A medication intake and administration record form will be provided to document the dose received and any adverse events reported by the participants. This form is designed to support adherence to the treatment regimen and serve as a "memory aid" to ensure compliance with therapy.

Inclusion criteria include: subjects of both sexes with primary, secondary or early latent syphilis. Exclusion criteria are: a) known allergy to any of the investigational drugs and/or excipients, in particular known hypersensitivity to penicillin, cephalosporin or other beta-lactam agents, b) clinical neurosyphilis, c) pregnant or lactating women, d) antibiotic treatment potentially active against T. pallidum (i.e., beta-lactams, cephalosporins, macrolides, tetracyclines) within the last week, e) concomitant symptomatic sexually transmitted disease (gonorrhea, chlamydia, lymphogranuloma venereum, Mycoplasma genitalium) or other infectious disease requiring antibiotic treatment potentially active against T. pallidum, f) having received treatment for syphilis.

The interventions planned to be performed on patients are as follows: clinical examination, blood count, hepatogram, renal function, urinalysis, serological studies (non-treponemal and treponemal test) for syphilis, qPCR for tpp47 gene of blood and/or lesions. And the laboratory parameters for the analysis are: kinetics of antibodies by RPR and Chemiluminescence. Paired (pre and posttreatment) qPCR results. Adverse events register per treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age up to 18 years.
2. Diagnosis of primary, secondary, or early latent syphilis, based on national and international standards (16, 17, 18).
3. Signed informed consent and assent.
4. Ability to comply with the study protocol requirements.
5. For women of childbearing potential, use of a highly effective contraceptive method (e.g., abstinence, hormonal contraception, or intrauterine device (IUD) is required. Contraception must be maintained for 1 week after the completion of treatment.
6. Male participants are advised to use condoms during sexual intercourse to prevent the transmission of syphilis to their partners.

Exclusion Criteria:

* 1. Known allergy or hypersensitivity to any of the investigational drugs or their excipients, particularly to penicillin, cephalosporins, or other beta-lactam agents.

  2. Diagnosis of clinical neurosyphilis. 3. Pregnant or lactating women. 4. Recent antibiotic treatment (within the past week) with drugs potentially active against Treponema pallidum, such as beta-lactams, cephalosporins, macrolides, or tetracyclines.

  5. Acute or chronic renal failure with a declining glomerular filtration rate. 6. Concomitant symptomatic sexually transmitted diseases (e.g., gonorrhea, chlamydia, lymphogranuloma venereum, Mycoplasma genitalium) or other infectious diseases requiring antibiotic treatment that could affect T. pallidum.

  7. Previous treatment for diagnosed syphilis. 8. Conditions that prevent oral administration of medication. 9. Other acute or chronic ailments or congenital disorders that, in the investigator's judgment, contraindicate participation in the trial or may interfere with the assessment of the efficacy, safety, or pharmacokinetics of the investigational product.

  10. Anticipated noncompliance with the protocol, treatment, or clinical trial testing and follow-up, as judged by the investigator.

  11. Cases involving prosecuted sexual abuse.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic Response Criteria | 2 weeks to 12 months
  •Serologic Response: An adequate serologic response is defined as a fourfold (2 dilutions) decrease in rapid plasma reagin (RPR) titer or seroconversion to a negative result during follow-up (6-12 months post-treatment).

SECONDARY OUTCOMES:
Adverse Events | 8 weeks
  Assessment of adverse events related to treatment with amoxicillin compared to those related to standard treatment with PGB within 8 weeks of treatment initiation.
Treatment Tolerance | 8 weeks
  Evaluation of treatment tolerance for amoxicillin versus PGB within 8 weeks of the start of the assigned treatment. The percentage of patients who do not complete treatment due to adverse events will be measured.
Antibiotic Response | 2 weeks to 12 months
  Evaluation of antibiotic response through the detection of negative Treponema pallidum (TPA) DNA by qPCR in paired samples (blood and swabs) collected before and after treatment during the scheduled visits

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Niños Ricardo Gutierrez, Buenos Aires City, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided